CLINICAL TRIAL: NCT06000956
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial Protocol of the Efficacy and Safety of Jitongning Tablets for Treating Spondyloarthritis (Kidney Yang Deficiency and Blood Stasis Obstruction)
Brief Title: A Study of Comparing Overall Improvement of Patients With Spondyloarthritis Treated With Jitongning Tablets and Placebo
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-JTNP-Ⅲ
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — jitongning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jitongning tablets (Experimental)
  Interventions: Drug: Jitongning tablets
- a simulated agent of Jitongning tablets (Placebo Comparator)
  Interventions: Drug: a simulated agent of Jitongning tablets

INTERVENTIONS:
Drug: Jitongning tablets — The participants took orally three tablets of Jitongning tablets, twice a day, for 8 consecutive weeks.
  Arms: Jitongning tablets
Drug: a simulated agent of Jitongning tablets — The participants took orally three tablets of a simulated agent of Jitongning tablets, twice a day, for 8 consecutive weeks.
  Arms: a simulated agent of Jitongning tablets

SUMMARY:
The goal of this clinical trial is evaluating the efficacy and safety of Jitongning tablets in participant population. The main questions it aims to answer are:

* Based on the proportion of participants who achieved improvement in ASAS20, evaluate whether the efficacy of Jitongning tablets is superior to placebo in active ax-SpA adult participants.
* Evaluate the efficacy of Jitongning tablets in improving other key functions and symptom outcomes.
* Evaluating the safety of Jitongning tablets in adult ax-SpA participants. Participants will

  1. take orally Jitongning tablets or a simulated agent of Jitongning tablets.
  2. Receive examinations and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

All of the following standards must be met:

1. Age range from 18 to 65 years old (including 18 and 65 years old), regardless of gender;
2. Meets the diagnostic criteria for axial osteoarthritis recommended by ASAS in 2009, and the condition is in an active phase. The criteria for determining disease activity are to meet two criteria: Bass ankylosing spondylitis disease activity index (BASDAI) ≥ 40mm (0-100mm, evaluated using VAS); Spinal pain score ≥ 40mm (0-100mm, evaluated using VAS);
3. Conforming to the traditional Chinese medicine syndrome differentiation standards for kidney yang deficiency and blood stasis obstruction syndrome;
4. CT examination of sacroiliac arthritis grades I (A) to II (B) (both included);
5. Human leukocyte antigen B27 (HLA-B27) is positive;
6. Elevated C-reactive protein (CRP)/hypersensitive C-reactive protein (hsCRP) and/or erythrocyte sedimentation rate (ESR);
7. Voluntarily participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

Those who meet any of the following criteria cannot be included in this experiment:

1. Received non-steroidal anti-inflammatory drugs within 2 weeks before enrollment;
2. Within 4 weeks before enrollment, he received traditional Chinese patent medicines and simple preparations or traditional Chinese medicine decoction, chemical drugs (such as sulfasalazine, methotrexate, leflunomide, hydroxychloroquine, cyclophosphamide, azathioprine, etc.), opioid analgesics (such as methadone, morphine, etc.), JAK inhibitor drugs (such as tofatib, etc.), and systemic glucocorticoid treatment;
3. Received spinal or joint surgery treatment within 8 weeks prior to enrollment;
4. Within 12 weeks prior to enrollment, biological agents with therapeutic effects on spinal arthritis have been used;
5. Within 6 months prior to enrollment, corticosteroid injections were received into the joint cavity or spine/paravertebral area;
6. CT indicates disappearance of sacroiliac joint space or complete spinal rigidity;
7. Subjects diagnosed with other rheumatic immune system diseases or immune deficiency syndrome, such as active ulcerative colitis, psoriasis, uveitis, etc;
8. Those who have fertility requirements within six months;
9. Pregnant or lactating women;
10. Suspected or actual drug, substance, or alcohol abuse;
11. Within 3 months prior to the trial or currently participating in clinical trials;
12. Serious heart, liver, kidney, brain, mental, and neurological disorders that affect informed consent and/or expression or observation of adverse events;
13. Abnormal liver function (elevated levels of alanine or alanine aminotransferase above the upper limit of normal values); Abnormal renal function (serum creatinine levels above the upper limit of normal values);
14. The researchers believe that it is not suitable to participate in this experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ASAS20 | 8 weeks
  Proportion of subjects who achieved improvement in ASAS20（Assessment of Spondylarthritis International Society） at week 8 of treatment.
  The ASAS Improvement Criteria contains the following 4 assessment domains:
  1. Physical function, by BASFI (Bath Ankylosing Spondylitis Functional Index);
  2. Spinal pain, by Spinal Pain Scale;
  3. Overall assessment of the condition in the past week, by PGA (Patient Global Assessment)
  4. Inflammatory activity, by the last 2 items of BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) were averaged.
  ASAS 20% response criteria (ASAS 20): 1. 3 of the above 4 items have at least ≥20% improvement and improved ≥ 10 mm in 0-100mm score; 2. Moreover, there was no deterioration in 1 item that did not achieve a 20% improvement from baseline.

SECONDARY OUTCOMES:
ASAS20 | 4 weeks
  Proportion of subjects who achieved improvement in ASAS20 at week 4 of treatment.The ASAS Improvement Criteria contains the following 4 assessment domains:
  1. Physical function, by BASFI (Bath Ankylosing Spondylitis Functional Index);
  2. Spinal pain, by Spinal Pain Scale;
  3. Overall assessment of the condition in the past week, by PGA (Patient Global Assessment)
  4. Inflammatory activity, by the last 2 items of BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) were averaged.
  ASAS 20% response criteria (ASAS 20): 1. 3 of the above 4 items have at least ≥20% improvement and improved ≥ 10 mm in 0-100mm score; 2. Moreover, there was no deterioration in 1 item that did not achieve a 20% improvement from baseline.
ASAS40 | 8 weeks
  Proportion of subjects who achieved improvement in ASAS40 at week 8 of treatment.The ASAS Improvement Criteria contains the following 4 assessment domains:
  1. Physical function, by BASFI (Bath Ankylosing Spondylitis Functional Index);
  2. Spinal pain, by Spinal Pain Scale;
  3. Overall assessment of the condition in the past week, by PGA (Patient Global Assessment)
  4. Inflammatory activity, by the last 2 items of BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) were averaged.
  ASAS 40% response standard (ASAS 40): 1. 3 of the above 4 items have at least ≥20% improvement and improved ≥ 20 mm in 0-100mm score; 2. Moreover, there was no deterioration in 1 item that did not achieve a 40% improvement from baseline.
spinal pain scale | 8 weeks
  Change from baseline in score of spinal pain at week 8 of treatment.The highest score on the scale is 100mm and the lowest is 0mm, and the higher the score, the more severe the condition.
BASFI | 8 weeks
  Change from baseline in score of BASFI（Bath Ankylosing Spondylitis Functional Index） at week 8 of treatment.The highest score on the scale is 100mm and the lowest is 0mm, and the higher the score, the more severe the condition.
PGA | 8 weeks
  Change from baseline in score of PGA（Patient Global Assessment） at week 8 of treatment.The highest score on the scale is 100mm and the lowest is 0mm, and the higher the score, the more severe the condition.
BASDAI | 8 weeks
  Change from baseline in score of BASDAI（Bath Ankylosing Spondylitis Disease Activity Index） at week 8 of treatment.The highest score on the scale is 100mm and the lowest is 0mm, and the higher the score, the more severe the condition.
Traditional Chinese medical Syndrome Points | 8 weeks
  Change from baseline in score of traditional Chinese medical Syndrome at week 8 of treatment.The scale has a maximum score of 36 points and a minimum score of 0 points, with lower scores indicating milder TCM symptoms.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Dongfang Hospital, Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Suzhou Hospital of Traditional Chinese Medicine, Suzhou, Jiangsu
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Yunnan Province Hospital of Traditional Chinese Medicine, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No